CLINICAL TRIAL: NCT04713878
Title: A 8-Week Trial of Mesenchymal Stem Cells Therapy in Patients With COVID-19 Pneumonia
Brief Title: Mesenchymal Stem Cells Therapy in Patients With COVID-19 Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayca Sultan Sahin, Assoc Prof, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.05.20
Record Dates: First submitted 2021-01-09; First posted 2021-01-19 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Coronavirus Disease 2019 (COVID-19) Pneumonia
Keywords: Mesenchymal stem cells; COVID-19; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Intervention Model Description: Coronavirus Disease 2019 (COVID-19) patients with pneumonia
  1.group: Intubated without comorbidity, 2.group: Intubated with comorbidity, 3.group: No intubated
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Intubated without comorbidity
  Interventions: Other: Mesenchymal stem cells
- Group 2 (Active Comparator): Intubated with comorbidity
  Interventions: Other: Mesenchymal stem cells
- Group 3 (Active Comparator): No intubated
  Interventions: Other: Mesenchymal stem cells

INTERVENTIONS:
Other: Mesenchymal stem cells — Intravenous infusion of Mesenchymal stem cells

SUMMARY:
Due to the cytokine storm that develops as a result of Coronavirus Disease 2019 (COVID-19) infection, some patients hospitalization to intensive care cause of pneumonia, Acute Respiratory Distress Syndrome (ARDS) and multiple organ failure. Mortality is higher in treatment-resistant cases.

Purpose of this study:

1. Providing immune modulation by Stem Cell Transplantation and reducing the damage caused by cytokine storm to tissues and organs,
2. Correcting immunosuppression and fight against COVID-19 virus by editing B and T cells,
3. It is to accelerate healing in organ damage by increasing growth factors through mesenchymal stem cells.

Primary outcome: Improvement of clinical symptoms, reduction of cytokine storm Secondary outcome: Recovery of patients; from mechanical ventilation

DETAILED DESCRIPTION:
Study design and participants This study was a single-center open-label, randomized trial conducted at an Education and Training Hospital, Istanbul from May to July, 2020, and it was performed according to the Declaration of Helsinki and approved by the Ethics Committee and health ministry (No:2020.05.20). Written informed consent was obtained from all patients or their representatives when data were collected prospectively.

Age, gender, mortality status, APACHE II score, number of days in ICU, procalcitonin and C-reactive protein values, leukocyte values, comorbid diseases, The cluster of differentiations 4 and 8 (CD4 and CD8), interleukin -2, interleukin -6, Tumor necrosis factor-alpha-beta levels will be recorded.

Clinical results, changes in inflammatory and immune function levels, and side effects will be recorded. The patient's lung function and symptoms will be recorded after Mesenchymal Stem Cell transplantation. After treatment, lymphocyte, C-reactive protein, Tumor Necrosis alpha-beta levels , interleukin-6 levels will be recorded.

Patients were divided into 3 groups:

1. group: Intubated without comorbidity (n:7)
2. group: Intubated with comorbidity (n:7)
3. group: No intubated (n:7)

Dosage of Mesenchymal stem cells:

1. 1 million cell/kg iv--------------------------------------------------day 0
2. 1 million cell/kg iv -------------------------------------------------day 2
3. 1 million cell/kg iv -------------------------------------------------day 4

ELIGIBILITY:
Inclusion Criteria:

* aged 18-90 male or female
* laboratory approve of RT-PCR (real-time reverse transcription polymerase chain reaction) with COVID-19 infection
* pneumonia assessed by chest radiography or computed tomography
* In accordance with any of the following: 1)Respiratory rate ≥ 30 times / min 2) oxygen saturation ≤ 93% 3) arterial pressure of oxygen/the fraction of inspired oxygen≤ 300mmHg, 4) pulmonary imaging of focus within 24-48 hours > 50% progression
* patients who remain unresponsive to medications administered according to Ministry of health guidelines
* Patients who receiving invasive or non-invasive mechanical ventilation therapy in intensive care

Exclusion Criteria:

* Pregnancy
* Any kind of cancer, severe liver disease
* Failure to provide informed consent or comply with test requirements
* Known allergy or hypersensitivity to MSCs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Change of clinical symptoms as respiratory distress or need for oxygen support | 3 months
  Recovery of patient from mechanical and oxygen support
Change of cytokine storm parameters | 3 months
  respiratory rates < 30 times /min
Change of pulmonary functions | 3 months
  Oxygen saturation > 93% and pulmonary imaging of focus within 24-48 hours > 50% progression
Change of clinical symptoms | 3 months
  arterial pressure of oxygen/the fraction of inspired oxygen>300mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Kaya, MD, Study Chair — Kanuni Sultan Suleyman Education and Training Hospital; Gursel Turgut, Prof Dr, Study Chair — Genkord; Ali Kocatas, MD, Study Chair — Kanuni Sultan Suleyman Education and Training Hospital
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT04713878/Prot_SAP_000.pdf